CLINICAL TRIAL: NCT06343103
Title: Multicentric Study to Evaluate Occupational Exposure to Antineoplastic Drugs Through Genotoxics Markers and Enviromental Monitoring
Brief Title: Study Evaluating Occupational Exposure to Antineoplastic Drugs
Acronym: BRIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEO 1735
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Cytotoxicity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workers exposed (Other): Workers exposed to cytotoxic agents
  Interventions: Other: Workers exposed
- Workers not exposed (Other): Workers not exposed to cytotoxic agents
  Interventions: Other: Workers not exposed

INTERVENTIONS:
Other: Workers exposed — Workers exposed to cytotoxic agents
  Arms: Workers exposed
Other: Workers not exposed — Workers not exposed to cytotoxic agents
  Arms: Workers not exposed

SUMMARY:
The multicenter study involves comparing two groups (an exposed group and a control group). The exposed group is selected from workers who perform their activities in drug handling areas (DH) or units for antineoplastic preparation (UFA), while the control group involves the voluntary participation of non-exposed workers (administrative staff).

The control group is selected based on the characteristics of the exposed group to ensure a homogeneous sample in terms of size and characteristics.

DETAILED DESCRIPTION:
The study will be proposed to all workers exposed to cytotoxic agents who have an employment contract or similar arrangement and who are affiliated with the hospital facilities participating in the protocol. Participation of workers in the study is voluntary.

The control group will be recruited from administrative staff and/or individuals not exposed to chemotherapy who have an employment contract or similar arrangement and who are affiliated with the hospital facilities participating in the protocol.

A subject is considered enrolled after signing the informed consent and will be considered evaluable if:

They have completed the exposure diary (only for the exposed group). They have responded to the medical history questionnaire. They have undergone sampling of oral mucosa exfoliated cells and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Capacity to understand and consent
* Personnel with an employment contract or similar arrangement
* Ability to comply with the procedures outlined in the protocol
* Signing of the informed consent

Exclusion Criteria:

* Age < 18 years old
* Any ongoing chemotherapy or radiation treatment for neoplasms of any kind
* Planned diagnostic exams involving radiation within three weeks following the signing of the Informed Consent
* Inability to comply with the procedures outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the difference in micronuclei frequency | 1 year
  Correlation between the difference in micronuclei frequency ain the exposed and unexposed groups

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Omodeo Salè, Principal Investigator — European Institute of Oncology
Locations (5):
- Italy (5):
  - IRCCS Ospedale Policlinico San Martino, Genova
  - European Institute of Oncology, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Napoli
  - Istituto Oncologico Veneto Irccs, Padua
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma